CLINICAL TRIAL: NCT06134882
Title: Smartphone-based Services for People Diagnosed With Opioid Use Disorder
Brief Title: OUD Smartphone Services
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Michigan University (Other)
Collaborators: DynamiCare Health Inc. (Unknown); RTI International (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB-2023-30; R44DA055396 (NIH)
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Opioid-Related Disorders; Drug Abuse
Keywords: Smartphone; Telemedicine; Motivation; Incentives; Contingency Management
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Investigators who have no direct contact with study participants will communicate directly with information technology (IT) staff to assign participants to one of the two study groups. Participants will be blind to hypothesis, and outcome assessors will be completely blind. Care providers (i.e., "Contingency Management [CM] Guides") cannot be blind because modified scripts are required for their interactions with participants depending on group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abstinence reinforcement (Experimental): Participants earn incentives for submission of salivary drug toxicology video selfies that show test results consistent with the goals of treatment. Goals are abstinence-based (i.e., relate to which tested substances should be negative on the test given the medications that the particular participant has been prescribed). Incentives are also provided for attendance at treatment-related appointments and for completion of self-paced cognitive behavior therapy modules available via the smartphone app.
  Interventions: Behavioral: Contingency management; Behavioral: Cognitive-Behavior Therapy Modules; Behavioral: Peer Contingency Management (CM) Guide
- Sample-contingent control (Sham Comparator): Identical to the experimental group except that incentives are available only for submission of selfie-videos that show test results, without regard to the results of the salivary drug toxicology test. Similarly, incentives are not provided for appointments or completion of wellness modules.
  Interventions: Behavioral: Drug testing; Behavioral: Wellness modules; Behavioral: Peer technical support

INTERVENTIONS:
Behavioral: Contingency management — Monetary incentives are delivered via reloadable debit card based on verified engagement in target behaviors, including drug abstinence, appointment attendance, and completion of self-paced cognitive behavior therapy modules.
  Other Names: Abstinence reinforcement
  Arms: Abstinence reinforcement
Behavioral: Cognitive-Behavior Therapy Modules — Self-paced cognitive-behavior therapy modules delivered via smartphone.
  Arms: Abstinence reinforcement
Behavioral: Peer Contingency Management (CM) Guide — Peer supports delivered via telehealth. Support is informed by the community reinforcement approach and includes motivational interviewing
  Arms: Abstinence reinforcement
Behavioral: Drug testing — Self-performed salivary drug testing with incentives contingent upon proper completion of test procedures as confirmed by video.
  Arms: Sample-contingent control
Behavioral: Wellness modules — Basic health and wellness information delivered via self-paced learning modules.
  Arms: Sample-contingent control
Behavioral: Peer technical support — Peer support for promoting engagement and addressing technical issues delivered via a mobile digital platform.
  Arms: Sample-contingent control

SUMMARY:
The purpose of the research is to check whether services and materials made available through a smartphone app are helpful to people who have been diagnosed with opioid use disorder (OUD). Participants are asked to use an app to submit videos of themselves taking salivary drug tests to a secure online system. The app includes reminders, rewards, and activities, as well as access to live support. Study participation lasts one year and includes about 30 minutes each week submitting videos, an hour-long interview to get started, and hour-long interviews once every three months after that over the course of the year.

DETAILED DESCRIPTION:
Purpose of the Study

The purpose of the study is to evaluate the safety, clinical effectiveness, and cost effectiveness of the standard DynamiCare Health smartphone-smartcard platform as a means of promoting health and recovery for patients who are seeking treatment for problem opioid use.

Experimental Design

This is a prospective parallel randomized controlled trial with two study arms. The experimental group receives a smartphone-based program that includes incentives contingent upon drug abstinence and treatment attendance, access to a contingency management (CM) Guide who provides measurement-based peer coaching grounded in Community Reinforcement Approach, and self-paced Cognitive Behavioral Therapy (CBT) modules. The control group receives a smartphone-based sham program that includes incentives for submission of self-conducted salivary toxicology tests.

Welcome Period

After recruitment, participants will complete the Welcome Period. Participants will earn a total of $67 for completing the Welcome Period after they have downloaded the app and enrolled.

After consenting, participants will enter the "Welcome" Period to learn the basics of how DynamiCare works before being randomized to a study condition. During the Welcome Period, participants will have their equipment shipped to them, attend an orientation, and earn rewards for completing non-contingent practice saliva tests. The practice tests will be pre-scheduled. Members will advance to study randomization once they have:

* Completed an enrollment call and provided informed consent ($10)
* Received their equipment in the mail (saliva test kits and debit card)
* Completed Orientation: A session to learn how to use the DynamiCare app and understand how to perform saliva testing ($10 reward)
* Completed initial required surveys: Brief Addiction Monitor ($2), Demographics ($5), and Quality of Life ($5)
* Completed 2 saliva tests ($5 reward each, $10 total) Participants will also earn a $25 bonus for completing the Welcome Period and accepting Randomization.

Randomization

Upon successful completion of the Welcome Period the DynamiCare study coordinator will notify the Western Michigan University (WMU) study coordinator that a participant randomization is required. The WMU study coordinator will notify the WMU principal investigator or WMU graduate student investigator who is scheduled as the randomizer that they should conduct the randomization as soon as possible. As part of this request, the WMU study coordinator must supply the answers to the three stratification questions.

The stratification variable questions are:

1. Do any salivary drug tests taken during the Welcome Period show use of unprescribed drugs [Y/N]?
2. Has the person been diagnosed with Stimulant Use Disorder or have problem stimulant use [Y/N]? and
3. Is the participant already enrolled in Medication for Opioid Use Disorder (MOUD) [Y/N]? Once randomization is complete, the randomizer will inform the WMU study coordinator, who will inform DynamiCare Enrollment Team staff in turn. The DynamiCare Enrollment Team will then ensure assignment to the appropriate condition and conduct a notification call. Note that the purpose of the notification call is to explain to the participant what will happen during their Study Period. UNDER NO CIRCUMSTANCE SHOULD THE PARTICIPANT BE TOLD WHETHER THEY ARE IN THE EXPERIMENTAL OR CONTROL CONDITIONS.

Once the participant is assigned to a condition in DynamiCare Analytics, they are considered fully enrolled and part of the intent-to-treat analysis.

Assessment Overview

Three types of assessments will be delivered throughout the study: Pre-Randomization, Self-Monitoring, and Major Assessments. A separate Excel file showing a diagram of all assessments and timepoints is available. This file also details the delivery mechanism and payment associated with each assessment.

* Pre-Randomization assessments will be delivered 1) either by phone during enrollment calls into the Welcome Period or 2) through the DynamiCare Health app during the Welcome Period before participants are randomly assigned to Study Period groups.
* Self-Monitoring assessments will be delivered through the DynamiCare Health app every 4 weeks throughout the study.
* Major Assessments will be delivered online and/or over the phone at five timepoints throughout the study. The exact schedule of all assessments is described in the subsections below.

Most importantly, all participants will receive identical assessments independent of their group assignment. The only exception to this is the "Invite a Supporter Survey." This assessment is delivered once to the experimental group only.

Interviews

Pre-Randomization Assessments.

1. American Society of Addiction Medicine (ASAM) Co-Triage (eligibility)
2. Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) Diagnostic Criteria Questionnaire (eligibility)
3. General Social Security Number Collection Form (enrollment call into Welcome Period)
4. Demographic Questionnaire (Welcome Period)
5. Brief Addiction Monitor (BAM) (Welcome Period)
6. The World Health Organization (WHO) Quality of Life (Welcome Period)

Self-Monitoring Surveys.

1. Brief Addiction Monitor (BAM) (intake and 4-week intervals)

Major Assessments.

1. Invite a Supporter Survey (intake for experimental group only)
2. WHO Quality of Life (intake/12-week intervals)
3. Delay and Probability Discounting Task (intake/24-week intervals)
4. Social Discounting Task (intake/24-week intervals)
5. Opioid Discounting and Purchasing Task (intake/24-week intervals)
6. Balloon Analog Risk Task (BART) (intake/24-week intervals)
7. Patient Health Questionnaire-9 (PHQ-9)
8. Timeline Followback (TLFB) for MOUD adherence (intake/12-week intervals intervals)
9. Treatment Status Questionnaire (intake/12-week intervals)
10. Economic Form 90 (EF90) Healthcare Utilization Questionnaire (intake and 12-week intervals)
11. Assessment of Blinding Success (12-week intervals excluding intake)
12. Satisfaction Survey (12-week intervals excluding intake)
13. Return to Work Self-Efficacy Survey (intake and 12-week intervals)
14. Flexpa data collection (intake, 24-week intervals)

Salivary Toxicology

Standard Salivary Toxicology. Salivary toxicology testing will be initially conducted twice per week, scheduled at random within the patient's designated time window (usually set between 8 AM-10 PM). For experimental group patients, the app uses a progressive reinforcement schedule for drug testing and rewards: with consecutive abstinences it tests the patient less frequently (e.g., eventually just every two weeks). With relapses, however, the app tests more frequently (e.g., up to two tests every week). The incentive amount is inversely related to the frequency of the tests, with a maximum of $30/week for all incentivized behavioral tasks (including CBT module completion and appointment attendance).

For the experimental group, substance tests will be reinforced contingent on abstinence from any non-prescribed drugs. A positive result for any prescribed drugs is not a requirement for reinforcement. For the control group, substance tests will be reinforced on a fixed schedule, contingent only on submission. All incentives will be available to participants through the 48-week Study Period.

The drug test panel that will be used with both study groups will include tests for a variety of opioids (e.g., including tests for buprenorphine, methadone, fentanyl), cocaine, methamphetamine, and benzodiazepines.

Primary Outcome Salivary Toxicology. In addition to the salivary drug toxicology tests that are performed according to the random schedule, there will also be a set of salivary toxicology tests that will be used as the primary outcome of the study. These tests will be independently analyzed by a laboratory at a frequency of once per month, with the first of these tests scheduled at the start of the Study Period. These samples will be sent to Quest Diagnostics for GC/Mass spec testing. A video selfie, sent to the WMU study team via OneDrive, will be required to ensure that the sample is properly provided by the correct participant. A payment of $20 will be made each month by the WMU study coordinator for the submission of this sample. Payment will be delivered after Quest Diagnostics provides the results of the toxicology test as confirmed by the WMU study coordinator.

Discharge Procedures

Main study discharge will occur for all participants irrespective of group assignment upon completion of the final assessment conducted on the 48th week of the study period.

Analytic Plan

All analyses will be conducted on the Intent-to-Treat population in SAS 9.3 or higher and all hypothesis testing will be two-sided with a 5% significance level (SAS Institute, Inc; Cary, NC, USA). Generalized Estimating Equations (GEE) and Mixed models will be used to evaluate all primary and secondary outcomes. The goodness of fit of the models will be assessed using the Quasi-likelihood under the Independence model Criterion (QIC) to choose the best-fitting correlation structure. For each model, effect sizes will be estimated as odds ratios (for binary outcomes), rate ratios (for count outcomes), or differences in means (for continuous outcomes). These estimates will be assessed for precision using 95% confidence intervals. Both GEE and Mixed statistical techniques are particularly suited for analyses of longitudinal data and allow for correlations among observations within an individual subject, for the presence of missing data, for subjects measured at different timepoints, and for covariates that change over time. The response of individual subjects is first modeled, and then the estimates for each individual are combined in a group analysis. These analyses will permit an examination for effects of assignment to treatment condition, time effects associated with the course of treatment, and condition by time interactions. Because the FDA considers people aged 18-21 to be adolescents, and people 22 or over to be adults, we will perform a sub-group analysis for adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Lives in the United States
* Read and speak English fluently
* Owns a smartphone compatible with the DynamiCare app (e.g., Apple or Android)
* Diagnosed with opioid use disorder or attests to having problem opioid use
* Has used unprescribed opioids within the prior 30 days
* Has, or is willing to accept, an appointment to initiate medication assisted treatment or has initiated medication assisted treatment in the prior 45 days
* Must have an ASAM CO-Triage score between L1 and L3.1

Exclusion Criteria:

* Is currently enrolled in another study involving substance abuse treatment
* Has concurrent alcohol use disorder
* Is currently incarcerated
* Has current suicidal ideation or overt psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Independent lab-based salivary drug toxicology for abstinence from all unprescribed drugs (initial 16 weeks) | Initial 16 weeks
  Abstinence from all unprescribed drugs as measured by independent, lab-based salivary toxicology testing (Y/N) collected every 4 weeks throughout the initial 16-week Study Period.

SECONDARY OUTCOMES:
Lab-based salivary drug toxicology for abstinence from all unprescribed drugs (weeks 17-48) | Weeks 17-48
  Abstinence from all unprescribed drugs as measured by independent, lab-based salivary toxicology testing (Y/N) collected every 4 weeks throughout weeks 17-48 of the Study Period, during which CM incentives have faded out in the experimental group as participants reach the CM earnings limit ($599).
Medications for Opioid Use Disorder (MOUD) participation | 48 weeks
  Self-reported MOUD participation status (Y/N) as assessed at quarterly assessments.
Days of Medications for Opioid Use Disorder (MOUD) adherence | 48 weeks
  Self-reported days of MOUD adherence as assessed at quarterly assessments.
Healthcare utilization | 48 weeks
  Healthcare utilization as assessed by the EF90 Healthcare Utilization Form. Assesses the following 90 days prior to completion:
  * Overnight stay (Y/N) in a hospital
  * Total nights spent in the hospital
  * Total nights spent in the hospital due to drugs, alcohol, or mental health
  * Overnight stay (Y/N) at treatment facility
  * Total nights spent in treatment facility
  * Emergency room visit (Y/N)
  * Total emergency room visits
  * Total emergency room visits related to alcohol, drug use, or mental health
  * Outpatient substance use disorder treatment or counseling (Y/N)
  * Total days of outpatient substance use disorder treatment or counseling
  * Use of medications to treat opioid use disorder (Y/N)
  * Total days of methadone use
  * Total days of buprenorphine use
  * Total injections of Vivitrol
Frequency of Adverse Events | 48 weeks
  Safety: Number of Adverse Events reported throughout the 48-week Study Period.

OTHER OUTCOMES:
Total Incentive earnings | 48 weeks
  Incentive earnings: Earning reported as a total and by category of behavioral target.
Self-reported drug use | 48 weeks
  Self-reported drug use (Y/N): Assessed as days of use in the past 30 days, as assessed every 4 weeks by the Brief Addiction Monitor (BAM).
Quality of Life assessment | 48 weeks
  Quality of Life as assessed every 12-weeks by the The World Health Organization Quality of Life (WHOQOL) survey. Each item of the assessment is scored from 1 to 5 from a five-point ordinal scale. The scores are then transformed linearly to a 0-100 scale with 0 representing the worst possible state of health and 100 indicating the best possible state of health.
Self-conducted abstinence from all unprescribed drugs | 16 weeks
  Abstinence from all unprescribed drugs as measured by self-conducted salivary drug toxicology testing (Y/N), through the DynamiCare app, collected weekly throughout the first 16 weeks of the Study Period, during which contingency management (CM) incentives will be included in the experimental group.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Michigan University, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Deposit complete deidentified data on openICPSR upon conclusion of the study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available upon approval of manuscript describing main study outcomes in a peer reviewed scientific journal. Data will remain on openICPSR indefinitely.
Access Criteria: Anyone.

DOCUMENTS (1):
  • Informed Consent Form (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT06134882/ICF_000.pdf